CLINICAL TRIAL: NCT04285008
Title: Randomized Controlled Study Comparing Colon Evaluation With The Pure-Vu System To A Standard Colonoscopy In Patients Who Are High Risk For Inadequate Bowel Preparation
Acronym: RESCue
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor has terminated study due to COVID-19 related concerns
Sponsor: Motus GI Medical Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: CL00048
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Gastrointestinal Disease; Colorectal Cancer
Keywords: colonoscopy
MeSH Terms: conditions — Gastrointestinal Diseases; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomization to Intervention or Control arm will use stratification by site, endoscopist and blocking. Sites are expected to contribute approximately equal numbers of procedures, and no site will be allowed to contribute more than 50% of the target sample size. The randomization sequences will be provided in advance by the study's statistician using an online system to obtain the randomization assignment and the corresponding colonoscope will be prepared. Randomization assignment will be recorded for each subject.
Who Masked: Participant
Masking Description: The Colonoscope will be prepared as per normal routine and the research assistant will cover the colonoscope before the patient enters the endoscopy room to keep him/her blinded to the study arm. This is uncovered once the patient is sedated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- standard Colonoscopy (No Intervention): Control arm
  Colonoscopy procedure using standard flushing and suctioning - standard of care
- Pure-Vu System (Other): Intervention - Colonoscopy procedure using Pure-Vu System
  Interventions: Device: Pure-Vu System

INTERVENTIONS:
Device: Pure-Vu System — The Pure-Vu System is Food and Drug Administration (FDA) approved device (K191220), intended to connect to standard colonoscopes to help facilitate intra-procedural cleaning of a poorly prepared colon by irrigating or cleaning the colon and evacuating the irrigation fluid (water), feces and other bodily fluids and matter, e.g. blood.
  Arms: Pure-Vu System

SUMMARY:
The primary objective of this multi-center, prospective, randomized controlled trial is to evaluate the bowel cleansing after Pure-Vu use in outpatient subjects at high risk for inadequate colon preparation as compare to standard of care.

DETAILED DESCRIPTION:
Total of 88 subjects (44 per arm) at high risk for inadequate colon preparation will be randomized and undergo procedure either in the Control arm (standard of care) or with the Pure-Vu System.

Subjects will be enrolled at up to 4 clinical sites in the United States.

primary endpoint- A comparison between the two study arms (i.e., Pure-Vu vs. standard colonoscopy) of the rate of overall cleansing as well as cleansing per segment will be evaluated by the BBPS scoring index (Bowel preparation adequacy defined as BBPS >2 in each segment)

The following secondary endpoints will be determined:

1. Assess the willingness of consented subjects to pay for Pure-Vu prior to colonoscopy
2. Colonoscopy procedural measures for Intervention and Control arms
3. Endoscopists' experience
4. Safety assessment for all subjects on the day of procedure per endoscopist
5. Post-colonoscopy patient experience and safety check with scripted phone call 1-3 days after colonoscopy
6. Assess the willingness of consented subjects to pay for the Pure-Vu System 1-3 days after colonoscopy

Follow-up call will be conducted 1-3 business days after the procedure to verify that there has been no change in their clinical status and record their willingness to use the Pure-Vu System in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Adults > age 22
2. Elective outpatient colonoscopy by participating gastroenterologist
3. Stool clarity grade 1-3 at presentation for colonoscopy

Exclusion Criteria:

1. Not competent to consent
2. Bleeding disorder - known or suspected
3. Hereditary Gastrointestinal Cancer syndrome
4. Known PT INR > 1.5
5. Know elevated PTT
6. Anti-platelet agent or anticoagulant (other than aspirin or nonsteroidal agent) which has not been stopped for the colonoscopy
7. Known platelet count < 50,000
8. Known absolute neutrophil count < 1,000
9. History of surgical colon resection
10. Pre-colonoscopy intent to enter terminal ileum
11. Prior incomplete colonoscopy due to technical & non-bowel preparation related reasons
12. Regular use of non-topical steroid
13. Pregnant
14. Prisoner or institutionalized for any reason
15. Psychiatric illness greater than mild
16. Colonoscopy without anesthesia administered (MAC) sedation
17. Diverticulitis
18. Active inflammatory bowel disease (Crohn's, Ulcerative Colitis, or Indeterminate)
19. Known or suspected colon stricture

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-04-15 (Estimated)

PRIMARY OUTCOMES:
rate of adequate cleansing level after using the Pure-Vu System as compare to sandard of care colonoscopy procedure | Up to 2 hours
  A comparison between the two study arms (i.e., Pure-Vu vs. standard colonoscopy) of the rate of overall cleansing as well as cleansing per segment will be evaluated by the BBPS scoring index (Bowel preparation adequacy defined as BBPS >2 in each segment)

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-12): https://cdn.clinicaltrials.gov/large-docs/08/NCT04285008/Prot_SAP_000.pdf